CLINICAL TRIAL: NCT02699957
Title: Left Atrial Appendage Occlusion Registry (LAAO Registry)
Status: Recruiting | Type: Observational
Sponsor: American College of Cardiology (Other)
Responsible Party: Sponsor
Other Study IDs: LAAO Registry
Record Dates: First submitted 2016-02-09; First posted 2016-03-07 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Atrial Fibrillation: Those patients with the condition of atrial fibrillation.
  Interventions: Procedure: Left Atrial Appendage Occlusion

INTERVENTIONS:
Procedure: Left Atrial Appendage Occlusion — Patients undergoing percutaneous/epicardial intervention for left atrial appendage occlusion.

SUMMARY:
The Left Atrial Appendage Occlusion Registry (LAAO Registry™) is designed to assess the prevalence, demographics, management, and outcomes of patients undergoing percutaneous and epicardial based left atrial appendage occlusion procedures to reduce the risk of stroke. Patient-level data will be submitted by participating hospitals on a quarterly basis to the American College of Cardiology Foundation's National Cardiovascular Data Registry (NCDR). The primary aims of the LAAO Registry are to optimize the outcomes and management of patients through the implementation of evidence-based guideline recommendations in clinical practice, facilitate efforts to improve the quality and safety for patients undergoing percutaneous and epicardial based left atrial appendage procedures, investigate novel quality improvement methods and provide risk-adjusted assessment of patients for comparison with nationwide NCDR data. The secondary purpose of the LAAO Registry is to serve as a rich source of clinical data to support assessments of short- and long-term safety, comparative and cost effectiveness research, and as a scalable data infrastructure for post market studies.

DETAILED DESCRIPTION:
Hospitals join the Left Atrial Appendage Occlusion Registry (LAAO Registry) by agreeing to the terms of a specific contract that outlines the obligations of each party and the annual fees for participation. In addition, participating sites sign a Business Associate Agreement with the American College of Cardiology (ACC) as per the requirements of the Health Insurance Portability and Accountability Act of 1996 (HIPAA).

The LAAO Registry dataset, comprised of approximately 300 data elements, was created by a panel of experts using available American College of Cardiology (ACC), Heart Rhythm Society (HRS), and Society for Cardiovascular Angiography and Interventions (SCAI) societal overview document guidance, data elements and definitions, previous trial data elements, and other evidentiary sources. Protected Health Information (PHI), such as social security number, is collected. The intent for collection of PHI is to allow for complete follow-up and tracking of the patient, to assist data managers in correcting data collection errors and improving data quality, for future registry interoperability and the potential for future generation of patient-level drill downs in Quality and Outcomes Reports (see section 11, Data Analysis and Statistical Considerations). Registry sites can opt out of transmitting direct identifiers to the National Cardiovascular Data Registry (NCDR), so inclusion of direct identifiers in the registry is at the discretion of the registry site. When using the NCDR web-based data collection tool, direct identifiers are entered but a partition between the data collection process and the data warehouse maintains the direct identifiers separate from the analysis datasets. The minimum level of PHI transmitted to the ACC when a participant opts out of submitting direct identifiers meets the definition of a Limited Dataset as such term is defined by the Health Insurance Portability and Accountability Act of 1996.

Data required for registry participation are collected retrospectively from existing medical records or concurrently in the normal course of treatment. The Societal Document and safety recommendations for left atrial appendage occlusion recommend additional testing and contact with the patient outside the hospital episode of care at 45 days, 6 months, 1 year and 2 years post-procedure. All registry data (in-hospital and follow-up) is captured by participating sites using an electronic data collection tool provided by the LAAO Registry or in the future the option will be available for collecting data using a certified software application that has been reviewed and certified as compliant with the transmissions specifications established by the ACC for the LAAO Registry.

Upon completion of a call for data window, participants prepare a data submission by exporting the data from their data collection mechanism and uploading their data to a secure https server at the ACC using approved encryption software with the highest encryption that is allowed.

In recognition of the importance of data quality to all of its registry products, and to ensure that data submitted to the NCDR are complete, consistent, and accurate, a Data Quality Program was formally established by the NCDR in 2004. Upon receipt of the LAAO Registry data submission, the ACC reviews the data electronically and reports back coding errors. Such electronic checks verify consistency and completeness and allow participants to have ample opportunity to submit data until it satisfies consistency and completion thresholds. The report produced from these data checks is called a Data Quality Report (DQR).

The DQR provides the participant with a confidential analysis of their data submission's completeness, and is used by the participant to help prioritize data cleaning efforts and to assess the necessity for re-submission.

Once the data meets the data quality thresholds, an Outcomes Report is produced. The Outcomes Report aggregates the participant's data and provides a comparison group (usually procedure volume based) and national comparison.

The NCDR understands the need to ensure the data submitted to the LAAO Registry is accurate and it has launched a national on-site and off-site audit program whereas a random set of participants participate in an on-site or off-site audit to confirm the data submitted to the registry is consistent with data in the medical record or source documentation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 years and older, undergoing percutaneous or epicardial left atrial appendage occlusion procedures

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All facilities performing percutaneous or epicardial left atrial appendage occlusion procedures.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-12; Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a major complication | Assessed in hospital for any occurence from the start of procedure date and time until discharge date and time, assessed up to 24 months. Reported quarterly.
  Proportion of patients experiencing any of the following events: Procedure aborted, conversion to open heart, hemorrhagic, ischemic or undetermined stroke, any effusion requiring drainage or surgery, device embolization, systemic embolism, or major bleeding event.

SECONDARY OUTCOMES:
Proportion of patients who experience a stroke (ischemic or hemorrhagic), or systemic embolism or death after left atrial appendage occlusion during the follow up timeframes | Assessed at 45 day, 6 month, 1 year and 2 year follow up
  Follow up metric for the proportion of patients who experience a stroke (ischemic or hemorrhagic), or systemic embolism or death after left atrial appendage occlusion.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Varosy, MD, Study Chair — VA Eastern Colorado Health Care System
Locations (1):
- American College of Cardiology/National Cardiovascular Data Registry (NCDR), Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: National Cardiovascular Data Registry (NCDR). Click this link for more information on the registry. — http://cvquality.acc.org
- Available data/document: Individual Participant Data Set: Data Collection Form — http://cvquality.acc.org/en/NCDR-Home/Data-Collection.aspx
- Available data/document: Individual Participant Data Set: Data Dictionary — http://cvquality.acc.org/en/NCDR-Home/Data-Collection.aspx — Element definitions and coding instructions.